CLINICAL TRIAL: NCT01420770
Title: A Phase 2 Randomized, Open-Label, Dose-Ranging Study of the Efficacy and Safety of Orally Administered SAR302503 in Patients With Intermediate-2 or High Risk Primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis, Post-Essential Thrombocythemia Myelofibrosis With Splenomegaly
Brief Title: Phase 2 Study of SAR302503 in Patients With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARD11936; U1111-1119-2965 (Other: UTN)
Record Dates: First submitted 2011-08-11; First posted 2011-08-22 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2016-02

CONDITIONS: Hematopoietic Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fedratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SAR02503 300 mg qd (Experimental): daily X 28 days
  Interventions: Drug: SAR302503
- SAR302503 400 mg qd (Experimental): daily X 28 days
  Interventions: Drug: SAR302503
- SAR302503 500 mg qd (Experimental): daily X 28 days
  Interventions: Drug: SAR302503

INTERVENTIONS:
Drug: SAR302503 — Pharmaceutical form:capsule
  Route of administration: oral

SUMMARY:
Primary Objective:

- To evaluate the efficacy of daily oral doses of 300 mg, 400 mg, and 500 mg SAR302503 for the reduction of spleen volume as determined by magnetic resonance imaging (MRI).

Secondary Objectives:

* To evaluate the safety of SAR302503.
* To evaluate the pharmacokinetics (PK) of SAR302503 after single and repeat doses.
* To evaluate the pharmacodynamics of SAR302503 as measured by changes in JAK2V617F allele burden in those patients with JAK2V617F mutation, changes in substrate phosphorylation in the JAK-STAT signal transduction pathway, and the expression of cytokines.
* To measure improvement in baseline Myeloproliferative Neoplasm (MPN) associated symptoms, as well as overall impact in quality of life (QOL), through serial administration of the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF).
* To measure generic health-related quality of life (HRQL) and utility values using the EQ-5D questionnaire.

DETAILED DESCRIPTION:
The duration of the study for an individual patient will include a period to assess eligibility (screening period 28 days), followed by a treatment period of at least 1 cycle (28 days) of study treatment, and an end-of-treatment visit at least 30 days following the last administration of study drug. However, treatment may continue if patients are deriving benefit and do not have unacceptable toxicity or meet study withdrawal criteria.

The study duration will be approximately 16 months which includes a 3-month enrollment period followed by a 12-month treatment period following the last patient enrolled followed by a 30-day follow-up period. The cut-off date for the analysis of the primary endpoint of response will be in maximum at the end of 3 months after the date of first dose of study drug of the last treated patient. The final analysis will be performed after the last enrolled patient completes the Cycle12 assessment.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of primary or post-polycythemia vera or post-essential thrombocythemia myelofibrosis (Post-ET MF) according to the 2008 World Health Organization (WHO) criteria
* Myelofibrosis classified as high-risk or intermediate-risk level 2, as defined by International Working Group - Myelofibrosis Research and Treatment (IWG-MRT)
* Enlarged spleen, palpable at least 5 cm below costal margin
* At least 18 years of age.
* Eastern Collaborative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2 at study entry.
* Adequate organ function
* Absence of active malignancy other than MF, except adequately treated basal cell carcinoma and squamous cell carcinoma of the skin, cervical carcinoma in situ or other malignancies that have been stable and off therapy for 5 years.
* Written informed consent to participate.
* Willing to comply with scheduled visits, treatment plans, laboratory assessments, and other study-related procedures.

Exclusion criteria:

* Splenectomy.
* Any chemotherapy (eg, hydroxyurea), immunomodulatory drug therapy (eg, thalidomide, interferon-alpha), immunosuppressive therapy, corticosteroids >10 mg/day prednisone or equivalent, or growth factor treatment (eg, erythropoietin), hormones (eg, androgens, danazol) within 14 days prior to initiation of study drug; darbepoetin use within 28 days prior to initiation of study drug.
* Major surgery therapy within 28 days or radiation within 6 months prior to initiation of study drug.
* Concomitant treatment with or use of pharmaceutical or herbal agents known to be at least moderate inhibitors or inducers Cytochrome P450 3A4 (CYP3A4), unless approved by the sponsor.
* Active acute infection requiring antibiotics.
* Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug.
* Participation in any study of an investigational agent (drug, biologic, device) within 30 days, unless during nontreatment phase.
* Prior treatment with a Janus kinase 2 (JAK 2) Inhibitor,
* Contraindications for undergoing Magnetic resonance imaging (MRI) (eg. metal implants).
* Pregnant or lactating female.
* Women of childbearing potential, unless using effective contraception while on study drug.
* Men who partner with a woman of childbearing potential, unless they agree to use effective contraception while on study drug.
* Known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness.
* Clinically active hepatitis B or C.
* Any severe acute or chronic medical, neurological, or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with interpretation of study results and, in the Investigator's opinion, would make the patient inappropriate for entry into this study.
* Unable to swallow capsules
* Presence of any gastric or other disorder that would inhibit absorption of oral medication.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The percent change in spleen volume based on MRI at the end of Cycle 3 relative to baseline | 1 year

SECONDARY OUTCOMES:
The proportion of patients who achieve ≥35% reduction in spleen volume from baseline, to Cycle 6 end of cycle (EOC) | 1 year
The percent change in spleen volume based on MRI at Cycle 6 EOC compared to baseline | 1 year
Duration of maintenance of ≥35% reduction in spleen volume relative to baseline, as measured at Cycle 3 EOC, at Cycle 6 EOC, after a year, after 18 months and after two years and at end of treatment (EOT). | 1 year
Characterization of the safety profile of SAR302503, including the frequency, duration, and severity of adverse events (AEs) 2 years | 1 year
Area under the plasma concentration versus time curve (AUC) of SAR302503 | 1 year
Peak plasma concentration (CMax) of SAR302503 | 1 year
In patients with the JAK2V617F mutation, change in peripheral blood granulocyte JAK2V617F allele burden from baseline to Cycle 3 EOC, to Cycle 6 EOC and at the end of every third cycle thereafter until Cycle 12 EOC and EOT | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- United States (4):
  - Investigational Site Number 840001, San Francisco, California
  - Investigational Site Number 840003, Ann Arbor, Michigan
  - Investigational Site Number 840006, Rochester, Minnesota
  - Investigational Site Number 840007, Canton, Ohio